CLINICAL TRIAL: NCT04558437
Title: Prevalence and Development of Post-traumatic Stress Disorder and Anxiety and Depressive Symptoms Among AP-HP Staff During the Covid-19 Epidemic
Brief Title: COVID-Impact "Psychological IMPACT of Covid-19 on AP-HP Staff"
Acronym: Covid-Impact
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: APHP200555
Record Dates: First submitted 2020-06-10; First posted 2020-09-22 (Actual); Last update posted 2020-09-22 (Actual); Status verified 2020-06

CONDITIONS: Post Traumatic Stress Disorder (PTSD); Anxiety; Depression; Epidemic Disease; COVID19
Keywords: prevalence; post-traumatic stress disorder (PTSD),; epidemic; COVID19
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Anxiety Disorders; Depression; COVID-19; Combat Disorders | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Questionnaire — Questionnaire at M0 M3 M6:
  PCL-5 (Post-Traumatic Stress Disorder Checklist Scale, version DSM-5) HAD (Hospital Anxiety and Depression Scale) SDS (Sheehan Disability Scales)

SUMMARY:
The epidemic of coronavirus induces a major influx of patients implying a rapid modification of the organizations, a work overload and a significant stress for the care teams and supports of the hospitals of the Assistance Publique - Hôpitaux de Paris (AP-HP) . To this is added the impact on each professional of the large number of very severe patients to be treated, of death and the anxiety of contamination, reinforced by the actual cases of staff themselves sick. Emergency phone numbers for professionals in the event of psychological suffering were quickly put in place at the AP-HP and Hospitals level. The objective of this study is to assess the psychopathological and psycho-traumatic consequences of this exceptional situation on the staff, during the epidemic and at a distance from it, in order to be able to target the solutions to be implemented. Hypothesis is that some personnel may develop one or more of the following disorders: adjustment disorder or other anxiety disorder, acute stress disorder, post-traumatic stress disorder (PTSD), and depressive episodes as defined in the DSM-5. This study also aimes to assess effect of support measures put in place, by comparing the evolution of those who benefited from those who did not use them, as well as the risk factors specific. The results will make it possible to have an estimate of the percentage of people who may require specific support, and to identify the staff most at risk, and thus predict the importance of the circuits and structures for support of staff which will be necessary in the short and long term. The main anticipated risk factors are: being a nurse, having a low number of years of professional experience, and being on the front line of care for affected patients.

ELIGIBILITY:
Inclusion Criteria:

* AP-HP professionals on duty during the COVID epidemic agreeing to participate in the three stages of the study.

Exclusion Criteria:

* none

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Care teams and supports of AP-HP hospitals
Sampling Method: Probability Sample
Enrollment: 20000 (Estimated)
Dates: Start 2020-06-12 (Actual); Primary Completion 2020-12-31 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Prevalence of PTSD among APHP staff during the COVID-19 epidemic and at a distance (inclusion, 3 months or 6 months). | 6 months
  Rate of respondents with a PTSD defined as score higher or equal to 32 for PCL-5 (Post-Traumatic Stress Disorder Checklist Scale, version DSM-5) at, at least, one of the three measures (inclusion, M3 or M6)

SECONDARY OUTCOMES:
Prevalence of Anxiety Disorder among APHP staff during the COVID-19 epidemic and at a distance (inclusion, 3 months and 6 months). | baseline, 3 months and 6 months
  Rate of respondents with an Anxiety Disorder defined as score higher or equal to 8 for the HAD-A subscale (Hospital Anxiety and Depression - Anxiety subscale) independently at each measure (inclusion, M3 and M6)
Prevalence of Depressive Disorder among APHP staff during the COVID-19 epidemic and at a distance (inclusion, M3 and M6). | baseline, 3 months and 6 months
  Rate of respondents with a Depressive Disorder defined as score higher or equal to 8 for the HAD-D subscale (Hospital Anxiety and Depression - Depression subscale) independently at each measure (inclusion, M3 and M6)

CONTACTS AND LOCATIONS:
Locations (1):
- Assistance Publique - Hôpitaux de Paris, Paris, Île-de-France Region, France

IPD SHARING:
Plan to Share IPD: No
DATAS ARE OWN BY ASSISTANCE PUBLIQUE - HOPITAUX DE PARIS, PLEASE CONTACT SPONSOR FOR FURTHER INFORMATION